CLINICAL TRIAL: NCT05840471
Title: Tranexamic Acid in Pregnant Women With Abruptio Placenta: A Double-blind, Multicenter Randomized Clinical Trial
Brief Title: Tranexamic Acid as an Intervention in Abruptio Placenta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, SHAHLA KAREEM ALALAF, Professor, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMU5
Record Dates: First submitted 2023-01-12; First posted 2023-05-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Vaginal Bleeding; Prolonged Pregnancy
Keywords: Abruptio placenta; Interventional study; Perinatal mortality; vaginal bleeding
MeSH Terms: conditions — Uterine Hemorrhage; Pregnancy, Prolonged; Abruptio Placentae; Perinatal Death | interventions — Tranexamic Acid; Glucose; Water

STUDY DESIGN:
Intervention Model Description: Randomization for both groups will be done using the Randomization Allocation Software program. Blindness in each group will be confirmed by a pharmacist who is not involved in the study and will have the codes belonging to the type of intervention with him until the end of the research.
  Random Allocation Software(https://random-allocation-software.software.informer.com/2.0/)
Who Masked: Participant, Investigator
Masking Description: Two similar size syringes will be prepared and labeled as A (experimental group) containing 1 g/10mL Tranexamic acid diluted with 20mL of 5% glucose water, and syringe B (placebo group) containing 30 mL of 5% glucose water.
  The 2 groups of syringes will be labeled with different numbers not known by the investigator or the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid group (Active Comparator): This interventional arm will receive tranexamic acid 1 g(10ml) (2 ampules each of 500 mg, 5ML) of tranexamic acid in 20 ml Dextrose 5% in water intravenously twice daily in the acute stage of bleeding for 48 hours. Participants will be followed up for recurrence of bleeding during pregnancy. The course of treatment will be repeated again if bleeding recurred. The hospital data safety and monitoring board ensured the continued safety of the Participants.
  Interventions: Drug: Tranexamic acid injection
- Dextrose 5% in water group (Placebo Comparator): Participants will receive 30 mL of Dextrose 5% in water slowly intravenously immediately during the attack of the bleeding, twice daily for 48 hours. Accompanied with the usual expectant management care.
  Interventions: Other: Dextrose 5% in water

INTERVENTIONS:
Drug: Tranexamic acid injection — This interventional arm will receive tranexamic acid 1 g (10ml) (2 ampules each of 500 mg, 5ML) of tranexamic acid in 20 ml Dextrose 5% in water intravenously twice daily in the acute stage of bleeding for 48 hours. Participants will be followed up for recurrence of bleeding during pregnancy. The course of treatment will be repeated again if bleeding recurred. The hospital data safety and monitoring board ensured the continued safety of the Participants.
  Other Names: Trenaxa; Macleods Pharmaceuticals Pvt.Ltd., Mumbai, India
  Arms: Tranexamic acid group
Other: Dextrose 5% in water — This interventional arm will receive tranexamic acid 1 g(10ml) (2 ampules each of 500 mg, 5ML) of tranexamic acid in 20 ml Dextrose 5% in water intravenously twice daily in the acute stage of bleeding for 48 hours. Participants will be followed up for recurrence of bleeding during pregnancy. The course of treatment will be repeated again if bleeding recurred. The hospital data safety and monitoring board ensured the continued safety of the Participants.
  Other Names: Glucose B.Braun
  Arms: Dextrose 5% in water group

SUMMARY:
Abruptio placenta is one of the common causes of antepartum haemorrhage which is more common in the second half of pregnancy and causes a high maternal and neonatal morbidity and mortality

DETAILED DESCRIPTION:
Abruption has been estimated to occur in 6.5 pregnancies per 1000 births, with an associated perinatal mortality rate of 119 per 1000 in the United States. A Cochrane database study revealed that there is no evidence from trials to show the best way to help pregnant women and their fetuses when there is a placental abruption. The baby may need to be delivered immediately, by cesarean section if alive, and often vaginally if the baby has died. Treatments include pain relief, blood transfusion, and monitoring. Bleeding during pregnancy is characterized by activation of the fibrinolytic system. Tranexamic acid is a potent pharmaceutical agent that suppresses fibrinolysis and thus can be used for managing hemorrhage in pregnancy. The FDA's pregnancy category for tranexamic acid is category B.

ELIGIBILITY:
Inclusion Criteria:

* 24 weeks gestation and more
* Stable hemodynamically
* Accepted to participate

Exclusion Criteria:

* Hypersensitivity to tranexamic acid
* Defective color vision
* History of venous thromboembolism
* Pre-existing medical conditions that could affect pregnancy outcomes (diabetes mellitus, hypertension, renal disease)
* Smoker
* Refused to participate in the trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Hemostasis | Up to time of delivery
  complete or gradual cessation of vaginal bleeding
Gestational age | at time of delivery
  37 weeks and more
Favorable perinatal outcome | up to 7 days post partum
  viable newborn, birth weight of at least 2,500 grams, an Apgar score of at least 7, and no neonatal intensive care unit hospitalization.
  more, birth weight of 2.5 kg and more

CONTACTS AND LOCATIONS:
Overall Officials: SHAHLA ALALAF, prof., Principal Investigator — Hawler Medical University
Locations (1):
- Shahla Kareem Alalaf, Erbil, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No
Will not be shared as is ethically unacceptable